CLINICAL TRIAL: NCT07010341
Title: Quantitative Intra-operative Assessment of Parathyroid Perfusion Using Indocyanine Green (ICG) Fluorescence Imaging: A Prospective Observational Study
Brief Title: Quantitative Intra-operative Assessment of Parathyroid Perfusion Using Indocyanine Green (ICG) Fluorescence Imaging
Status: Recruiting | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Bo Wang,MD, Director, Head of Thyroid Surgery, Principal Investigator, Clinical Professor, Fujian Medical University
Other Study IDs: PT-ICG
Record Dates: First submitted 2025-05-25; First posted 2025-06-08 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-05

CONDITIONS: Thyroid Surgery
Keywords: Thyroid surgery; Indocyanine Green; Near-Infrared Fluorescence; Parathyroid Perfusion; Perfusion Threshold; Hypocalcemia; Perfusion Ratio
MeSH Terms: conditions — Hypocalcemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Derivation_Cohort: The model-development cohort consisted of 500 consecutive patients drawn from the Thyroid Surgery Department database of Fujian Medical University Union Hospital (Fuzhou, China)
  Interventions: Diagnostic Test: ntra-operative Indocyanine Green (ICG) Fluorescence Quantification
- Validation_Cohort: The external validation cohort comprised 300 patients
  Interventions: Diagnostic Test: ntra-operative Indocyanine Green (ICG) Fluorescence Quantification

INTERVENTIONS:
Diagnostic Test: ntra-operative Indocyanine Green (ICG) Fluorescence Quantification — After a single intravenous bolus of indocyanine green (25 µg/kg), a near-infrared sensor records raw fluorescence intensity from the superior parathyroid gland and the ipsilateral common carotid artery at 60-120 seconds. No images are stored; only peak intensity values are logged to calculate the perfusion ratio R = PTG / CCA. The measurement is observational, adds ≤2 minutes to operative time, and involves no therapeutic intent.

SUMMARY:
This single-center, prospective, three-phase observational cohort quantifies the relationship between indocyanine green (ICG) fluorescence and early parathyroid function. Adult patients scheduled for unilateral thyroid lobectomy with autotransplantation of the ipsilateral inferior parathyroid gland are enrolled. After intravenous ICG 25 µg/kg, peak fluorescence of the superior parathyroid gland and the common carotid artery (CCA) is recorded at 60-120 seconds to calculate the ratio R = PTG/CCA. Serum parathyroid hormone (PTH) is measured 30 minutes post-operatively. A derivation cohort (~120 patients) generates R-based thresholds for in-situ preservation versus autotransplantation, which are prospectively validated in an independent cohort (60 patients) together with decision-curve analysis of clinical net benefit.

DETAILED DESCRIPTION:
Post-thyroidectomy hypocalcemia, reported in 5-30 % of cases, is largely attributable to inaccurate assessment of parathyroid perfusion. Conventional intra-operative judgment-based on gland color, capillary bleeding and pulsation-is subjective and non-quantitative. Near-infrared fluorescence imaging with indocyanine green (ICG) allows real-time visualization of tissue perfusion, yet no widely accepted quantitative threshold exists to guide in-situ preservation versus autotransplantation of parathyroid glands.

The PT-ICG study addresses this gap through:

Target population: Patients undergoing unilateral thyroid lobectomy with planned autotransplantation of the ipsilateral inferior parathyroid gland, isolating evaluation to the superior gland.

Pilot phase (n=30): Optimization confirmed an ICG dose of 25 µg/kg and a 60-120 s acquisition window, with the common carotid artery (CCA) providing a stable reference; well-perfused glands exhibited R values ~0.8-3.0.

Derivation phase (n≈120): The relationship between R and 30-min postoperative PTH is modeled; ROC analysis and the Youden index yield R_low and R_high thresholds, internally validated with bootstrap resampling.

Validation phase (n=60): Prospective application of thresholds documents surgeon decisions, postoperative PTH, and hypocalcemia incidence; predictive performance (AUC, sensitivity, specificity) and net clinical benefit (decision-curve analysis) of the R-based strategy are compared with standard clinical judgment.

Sample size and statistics: With an anticipated correlation r≈0.45, α=0.05 (two-sided) and 90 % power, ≥110 patients are required; allowing 10 % attrition, 120-130 will be enrolled.

Data management and safety: REDCap will support double data entry and monitoring; ICG-related adverse events will be recorded; the study adheres to GCP and the Declaration of Helsinki and has received ethics committee approval.

By establishing actionable ICG fluorescence thresholds and a decision algorithm, the study seeks to provide a quantitative tool for real-time intra-operative perfusion assessment, potentially reducing hypocalcemia and informing future multicenter trials.

full SAP available upon request / will be posted as separate document.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for unilateral thyroid lobectomy plus central (VI-level) lymph-node dissection.
* Intra-operative findings consistent with:
* Complete identification and in-situ preservation of the ipsilateral superior parathyroid gland;
* Complete identification and autotransplantation of the ipsilateral inferior parathyroid gland.
* Serum 25-hydroxy-vitamin D ≥ 30 ng/mL at baseline; patients below this level may be enrolled after standardized vitamin-D and calcium supplementation with re-test confirming ≥ 30 ng/mL.
* Surgery and all postoperative follow-up performed at the study center.
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Prior surgery on the thyroid or parathyroid glands.
* Severe hepatic or renal impairment, or other serious metabolic bone disease.
* Pregnancy or lactation.
* Known hypersensitivity to indocyanine green or iodine-containing compounds.
* Inability or unwillingness to comply with postoperative visits and blood testing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive adult patients undergoing unilateral thyroid lobectomy with planned autotransplantation of the ipsilateral inferior parathyroid gland at a single tertiary endocrine-surgery center; recruitment limited to cases in which the superior parathyroid gland can be preserved in situ and evaluated intra-operatively with indocyanine-green fluorescence quantification.
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Parathyroid Gland Fluorescence Intensity | Intra-operative (60 - 120 s post-ICG)
  Peak fluorescence intensity of the ipsilateral superior parathyroid gland, captured 60 - 120 seconds after a single intravenous bolus of indocyanine green (25 µg/kg).
Common Carotid Artery (CCA) Fluorescence Intensity | Intra-operative (60 - 120 s post-ICG)
  Peak fluorescence intensity of the ipsilateral common carotid artery recorded in the same 60 - 120 second window; serves as the reference signal for perfusion ratio calculations.
Parathyroid Hormone (PTH) at 30 Minutes post-surgery | 30 minutes after surgery
  PTH concentration (pg/mL) measured by chemiluminescent assay 30 minutes after skin closure, reflecting immediate functional status of the preserved superior parathyroid gland.

SECONDARY OUTCOMES:
Administered ICG Dose | Intra-operative (time of injection)
  Total dose of indocyanine green (µg/kg) delivered during the procedure.
PTH at 6 Hours | 6 hours post-surgery
  PTH concentration measured 6 hours after surgery.
PTH at 2 Weeks | 2 weeks post-surgery
  PTH concentration measured 14 ± 2 days after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided